CLINICAL TRIAL: NCT01040247
Title: Optimal Timing For Embryo Transfer For Low Responder Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amir Weiss, Senior Physician, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0027-09-EMC
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
Keywords: Infertility; Low Responder; IVF; Embryo Transfer
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

ARMS (2):
- Day 0 Embryo Transfer (Experimental): Embryo transfer will be performed on the same day as oocyte aspiration and fertilization
  Interventions: Other: Embryo Transfer
- Day 2,3 Embryo Transfer (Active Comparator): Embryo Transfer will be performed 2 or 3 days after oocyte aspiration and fertilization
  Interventions: Other: Embryo Transfer

INTERVENTIONS:
Other: Embryo Transfer — In the study group embryo transfer will be performed on the day of oocyte aspiration and fertilization while in the control group it will be done 2 or 3 days later as is common practice.

SUMMARY:
Women undergoing in vitro fertilization (IVF) therapy, who are low responder and agree to enter the trial will be randomized to a study group, for whom embryo transfer will be done on the same day as oocyte aspiration and fertilization; and a control group for whom embryo transfer will be performed 48 to 72 hours later, as is the current accepted practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing IVF
* Number of mature oocytes equal to or lesser than the maximum number of embryos intended for transfer

Exclusion Criteria:

* Patient nor consenting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel